CLINICAL TRIAL: NCT01648088
Title: Enhanced Detection of Staphylococcus Aureus Colonization in Patients Undergoing Prosthetic Joint Implantation.
Brief Title: Detection of Staph Colonization in Pre-op Arthroplasty Patients
Acronym: Staph
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0569-11-EP
Record Dates: First submitted 2012-06-28; First posted 2012-07-24 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Surgical Site Infection
Keywords: staphylococcus aureus; prosthetic joint implantation
MeSH Terms: conditions — Surgical Wound Infection; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-op THA and TKA patients: Patients who are scheduled for total joint arthroplasty

SUMMARY:
This study will evaluate which body site(s) provide the best source of possible staph presence in participants undergoing total joint arthroplasty. If the pre-operative cultures indicate staph presence, an Infectious Disease specialist will be consulted for standard of medical care consultation and treatment management. Participants will be followed for 2 years post-implantation of prosthetic joint to monitor development of prosthetic joint infection.

DETAILED DESCRIPTION:
The presence of Staph in/on a patient who will undergo total joint replacement is a risk in that the patient could go on to develop infection at the surgery site after surgery. The purpose of this study is to evaluate if it is beneficial to to administer a questionnaire and obtain cultures from various body sites from patients prior to surgery and also to determine which body site(s) provide the best source of possible staph presence. If the pre operative cultures indicate staph is present, an Infectious Disease specialist will be consulted for standard of medical care consultation and treatment management. All patients scheduled to have total joint arthroplasty are eligible to participate. The research team will follow the study patients for 2 years after they undergo prosthetic joint implantation to monitor for development of prosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing prosthetic joint implantation

Exclusion Criteria:

* None

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing prosthetic joint implantation.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Development of surgical site infection. | Change in surgical site from baseline at 6 months, 1 year, 18 months and 2 years.
  The patient will be assessed by phone every 6 months for 2 years for development of infection at the surgical site.

SECONDARY OUTCOMES:
Anatomical site(s) which are best utilized for swab cultures to detect S aureus. | Up to 24 months post operatively.
  We hope to determine which anatomical site(s) are best utilized for swab cultures to detect S aureus colonization in patients undergoing prosthetic joint replacement. We will collect data on infection development for up to 2 years post operatively.
Post operative infection (s.aureus) development. | Up to 24 months post operation.
  We will measure at what percentage a pre-operative questionnaire accurately predicts if a patient will develop an infection (s.aureus) between day one and 2 years post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hewlett, MD, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States